CLINICAL TRIAL: NCT06201390
Title: Effect of Stable Sleep Patterns on Peripheral Vascular Function Following Sleep Deprivation
Brief Title: Stable Sleep Pattern Before Sleep Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Joaquin U Gonzales, PhD, Associate Professor, Texas Tech University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB2023-1166
Record Dates: First submitted 2023-12-14; First posted 2024-01-11 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Sleep
Keywords: sleep variability; blood pressure; sleep deprivation; vasodilation
MeSH Terms: conditions — Sleep Deprivation; Aneurysm

STUDY DESIGN:
Intervention Model Description: Participants will complete a 6-week study that will involve five study visits. The first visit will include informed consent, collection of demographic data, sleep- and health-related surveys, and familiarization with study procedures. Participants will then be block randomized to either habitual sleep followed by stable sleep, or stable sleep followed by habitual sleep - each sleep condition will lasts two weeks. In the habitual sleep condition, participants will be asked to follow their normal routine without concern about their sleep duration. In the stable sleep condition, participants will be asked to keep the same bedtime and wake-time schedule without deviation. Blood pressure, blood vessel vasodilatory function, and cardiovascular responses to exercise will be our main outcome variables. These variables will be measured before (on day #13) and after (on day #14) one night of sleep deprivation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stable sleep (Experimental): Participants will be asked to maintain a consistent sleep pattern for two weeks.
  Interventions: Behavioral: Sleep consistency
- Habitual Sleep (No Intervention): Participants will be asked to maintain their usual sleep pattern for two weeks.

INTERVENTIONS:
Behavioral: Sleep consistency — Participants will be asked to maintain a consistent bed- and wake-time.
  Arms: Stable sleep

SUMMARY:
Sleep is now recognized as important for disease prevention. Too little or too much sleep contributes to cardiovascular disease. Leading health organizations recommend adults sleep 7-9 hours per night for optimal health. This recommendation is based on research that finds reductions in sleep duration elevate blood pressure and impair vasodilation of blood vessels. One question raised in a recent NIH Workshop report (PMID:36448463) is whether stable sleep patterns, irrespective of a person's sleep duration, could mitigate the adverse effects of insufficient sleep on vascular function. This project will address this question in midlife adults using a randomized, crossover designed study.

DETAILED DESCRIPTION:
Purpose and hypothesis The aim of this study will be to test the hypothesis that stable sleep, as defined by a consistent (low variability) bedtime and wake-time schedule, will diminish the negative effect of sleep deprivation on vascular function.

Study design and procedures Thirty adults (15 men, 15 women) will complete a 6-week study that will involve five study visits. The first visit will include informed consent, collection of demographic data, sleep- and health-related surveys, and familiarization with study procedures. Participants will then be block randomized to either habitual sleep followed by stable sleep, or stable sleep followed by habitual sleep - each sleep condition will lasts two weeks. In the habitual sleep condition, participants will be asked to follow their normal routine without concern about their sleep duration. In the stable sleep condition, participants will be asked to keep the same bedtime and wake-time schedule without deviation. Bedtime and wake-times will be determined by the researchers, but individualized for each participant so that their usual sleep duration (based on self-report) is met. Sleep will be monitored throughout the study using research-grade motion sensors worn at the wrist. Resting blood pressure, blood vessel vasodilatory function, and cardiovascular responses to exercise will be our main outcome variables. These variables will be measured before (on day #13) and after (on day #14) one night of sleep deprivation. Total sleep deprivation is a well-established experimental model to understand the acute effects of insufficient sleep on vascular function in humans.

ELIGIBILITY:
Inclusion Criteria:

* Women and men
* 35-64 years of age

Exclusion Criteria:

* obese based on BMI >29 kg/m2
* night-shift work
* prior diagnosis of sleep apnea
* signs of insomnia using the Insomnia Symptom Questionnaire
* a 'poor sleeper' (global score ≥5) based on the Pittsburgh Sleep Quality Index
* taking medications that alter sleep
* personal history of stroke, coronary heart disease, diabetes mellitus
* taking antihypertensive medications
* smoker (including vaping)

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-02-08 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Change in Peak Reactive Hyperemia | pre-intervention; immediately after the intervention
  Peak forearm blood flow will be measured before and after one night of sleep deprivation that follows two weeks of normal sleep or stable sleep. Peak reactive hyperemia in the forearm (ml/100ml/min) will be measured using venous occlusion plethysmography after 10 minutes of forearm ischemia resulting from blood pressure cuff inflation at the upper-arm. Peak blood flow is considered the highest blood flow measurement after the blood pressure cuff is deflated.
Change in Arterial Stiffness | pre-intervention; immediately after the intervention
  Arterial stiffness will be measured measured before and after one night of sleep deprivation that follows two weeks of normal sleep or stable sleep. Carotid-femoral pulse wave velocity will be used as the measure of arterial stiffness. Radial arterial tonometry will be used to derive a central aortic blood pressure wave. Wave separation analysis of the aortic pressure wave will then used to calculate pulse wave velocity from transit time and carotid-femoral path length.
Change in Blood Pressure Reactivity | pre-intervention; immediately after the intervention
  Blood pressure responses to isometric handgrip exercise will be measured before and after one night of sleep deprivation that follows two weeks of normal sleep or stable sleep. Mean blood pressure reactivity will be measured using finger plethysmography during 2-minutes of isometric handgrip exercise followed by 3-minutes of post-exercise circulatory arrest.
Change in Cerebral oxygenation | pre-intervention; immediately after the intervention
  Regional cerebral oxygenation during a cognitive task will be measured before and after one night of sleep deprivation that follows two weeks of normal sleep or stable sleep. Oxy- and deoxy-hemoglobin levels in the prefrontal cortex will be measured using a near infrared spectroscopy (NIRs) device.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin U Gonzales, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Kinesiology and Sport Management building, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All data collected or generated from the project will be made available on ClinicalTrials.gov within 12 months from the primary completion date.
Supporting Information: ICF
Time Frame: All data collected or generated from the project will be made available on ClinicalTrials.gov within 12 months from the primary completion date.
Access Criteria: Open access

DOCUMENTS (1):
  • Informed Consent Form (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT06201390/ICF_000.pdf